CLINICAL TRIAL: NCT01503320
Title: Efficacy of Enteral Glutamine Supplementation in Patients With Predicted Severe Acute Pancreatitis- A Double-Blinded Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: AIG-GI-2011-05
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Acute Pancreatitis
Keywords: To evaluate; efficacy; enteral glutamine
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enteral glutamine (Experimental)
  Interventions: Dietary Supplement: Enteral glutamine
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Enteral glutamine — Dosage of glutamine: 0.57g/kg, ~ 30g/day= 3sachets
  Arms: Enteral glutamine
Dietary Supplement: Placebo — Similar appearing nutritional supplement without glutamine.
  Arms: Placebo

SUMMARY:
Acute pancreatitis (AP) is a potentially serious illness characterized by inflammation of the pancreas with variable involvement of peri-pancreatic tissues and/ or remote organ systems. AP is hyper catabolic condition due to systemic inflammatory response syndrome (SIRS without any proven specific treatments. Therefore, current therapy for AP is directed to intensive medical care, nutrition support and infection control.

Nutritional support is very crucial in the treatment of AP. Enteral nutrition (EN) is the preferred modality since parenteral nutrition is associated with various complications. EN could preserve the intestinal permeability, which would be the best barrier for prevention of certain complications.

Glutamine is the most abundant free amino acid in the body and is used as a major fuel and nucleotide substrate. When a nutritional deficiency arises in critical illness including SAP, glutamine tends to be conditionally depleted.

We hypothesize that enteral glutamine supplementation in patients with severe and predicted severe acute pancreatitis helps in their early recovery and prevention of adverse outcomes.

In this study, we aim to evaluate the therapeutic effect of enteral glutamine on clinical outcomes, gut permeability, systemic inflammation, oxidative stress and plasma glutamine levels.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a potentially serious illness characterized by inflammation of the pancreas with variable involvement of peri-pancreatic tissues and/ or remote organ systems. AP contributes to thousands of annual hospital admissions, of which severe acute pancreatitis (SAP) accounts for 10-20%. The course of SAP tends to be prolonged and the patients usually are hyper metabolic and high protein catabolic due to systemic inflammatory response syndrome (SIRS) induced by acute local inflammatory process and subsequent vital organ dysfunction. There are currently no specific proven treatments. Therefore, current therapy for AP is directed to intensive medical care, nutrition support, infection control and medicine administration.

Nutritional support plays an important role in the management of patients with SAP, which is very critical and complex. Thus, if nutritional support is not appropriately administered to match the rapidly increasing demand in the treatment of SAP, the patients consequently come down with gross metabolic imbalance and nutrition deficiency. This is considered to increase mortality due to impaired immune function, increased risk of infections and intractable vital- organ failure.

Despite the recently reported encouraging results on early enteral feeding in patients with acute pancreatitis, total parenteral nutrition (TPN) is still frequently performed in the management of patients with AP. However, longer periods of TPN are known to be associated with mucosal atrophy and increased gastrointestinal permeability, two established risk factors for endotoxemia and bacteriemia.

Artificial nutrition can prevent complications and provide long term nutritional support for SAP patients. Enteral nutrition is preferred to parenteral nutrition for improving patient outcomes and has largely replaced the parenteral route. Early nasogastric enteral nutrition (NGEN) was considered potentially to lead to pancreatic-unrest and thereby prove to be harmful to the early acute phase of AP. However, Eatock et al introduced the early nasogastric feeding into the nutritional management of SAP and Pandey et al applied oral re-feeding in patients with SAP, suggesting that the nasogastric feeding is feasible in up to 80% cases. A meta-analysis and a recent randomized controlled trial showed that early NGEN would be as effective and safe as early Naso Jejunal enteral nutrition (NJEN) or TPN in SAP patients, without increase in mortality and pain on re-feeding.

EN could preserve the intestinal permeability, proven by the assessment of excretion of polyethylene glycol and antiendotoxin core antibody IgM levels, which would be the best barrier for prevention of certain complications. Serum interleukin-6 levels are elevated very early in patients with necrosis infection and C-reactive protein (CRP) is considered a valuable independent predictor of mortality. IL-6 and CRP levels play a similar role in the control of systematic inflammatory response of early EN and TPN groups at each time point. Moreover, biochemical/ nutritional parameters such as serum albumin and prealbumin concentration in early EN are well preserved without any significant difference.

Glutamine is the most abundant free amino acid in the body. When a nutritional deficiency arises in critical illness including SAP, glutamine, readily synthesized under most situations, tends to be conditionally depleted. The low concentration of plasma glutamine was found to be an independent predictive factor for a poor outcome in critical illness. Glutamine is used as a major fuel and nucleotide substrate for rapidly dividing cells such as intestinal mucosal cells and the gut-associated immunocytes. Glutamine can prevent atrophy of the intestinal epithelial cells through HSP 70 generation and improve the intestinal immune barrier. A meta-analysis by Novak et al revealed that glutamine could reduce the infectious morbidity (RR 0.84, 95% CI: 0.68-1.03) and mortality (RR 0.76, 95% CI: 0.56-0.98) in critical illness.

Standard TPN does not contain glutamine. Parenteral nutrition supplemented with glutamine showed a beneficial effect on preservation of the intestinal integrity, improving lymphocyte function and improving antioxidant capacity compared to a standard TPN; and glutamine administration was related to a clinically significant decrease in morbidity and mortality.

We hypothesize that enteral glutamine supplementation in patients with severe and predicted severe acute pancreatitis helps in their early recovery and prevention of adverse outcomes.

In this study, we aim to evaluate the therapeutic effect of enteral glutamine on clinical outcomes, gut permeability, systemic inflammation, oxidative stress and plasma glutamine levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age 18.
* Patient admitted within 72hrs of onset of abdominal pain for over 24hr with raised (>3- fold) serum lipase/amylase on admission.
* Marshall Score of ≥ 2 in any one organ, excluding the liver component
* Pancreatic necrosis >30% on Computed tomography (CT) scan or a modified CT severity index of ≥6.
* Apache II score ≥8.
* BUN at admission of >20mg/dL or an BUN elevation of >5mg/dL within 48hrs of admission.

Exclusion Criteria:

* Patients with chronic pancreatitis and pancreatic insufficiency requiring pancreatic enzyme supplements.
* Pre-existing chronic renal insufficiency requiring hemodialysis or peritoneal dialysis.
* Patients with ARF.
* Pre-existing end-stage liver disease with ascites, coagulopathy and encephalopathy.
* Pancreatic cancer.
* Current somatostatin or corticosteroid therapy.
* Any form of artificial feeding since commencement of acute pancreatitis symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Development of infected (peri)pancreatic necrosis | Baseline; 7 days; 6 months
Mortality | Baseline; 7 days; 6 months

SECONDARY OUTCOMES:
Change in levels of HS- CRP. | Baseline, 7 days, 14 days
Change in mucosal permeability | Baseline, 7 days, 14 days
Change in level of oxidative stress | Baseline, 7 days, 14 days
Change in cytokine levels in serum | Baseline, 7 days, 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Rupjyoti Talukdar, MD, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India

REFERENCES:
- [Derived] Arutla M, Raghunath M, Deepika G, Jakkampudi A, Murthy HVV, Rao GV, Reddy DN, Talukdar R. Efficacy of enteral glutamine supplementation in patients with severe and predicted severe acute pancreatitis- A randomized controlled trial. Indian J Gastroenterol. 2019 Aug;38(4):338-347. doi: 10.1007/s12664-019-00962-7. Epub 2019 Oct 14. PMID 31612309